CLINICAL TRIAL: NCT02224612
Title: A Comparative Evaluation of the Performance and Fit of Pediatric Face Masks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R13-044
Record Dates: First submitted 2014-01-08; First posted 2014-08-25 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Pediatric Face Masks; children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Children 4-5 yrs (Active Comparator): Medline Pediatric Face Mask KC Childs Face Mask
  Comparison of Medline Pediatric Face Masks and KC Childs Mask which are both single use disposable masks. Each mask (two in total) were worn for 2-3 minutes for EtCO2 and respiration assessments and physical fit assessment.
  Interventions: Device: Medline Pediatric Face Masks; Device: KC Childs Mask
- Children 6-9 yrs (Active Comparator): Medline Pediatric Face Mask KC Childs Face Mask
  Comparison of Medline Pediatric Face Masks and KC Childs Mask which are both single use disposable masks. Each mask (two in total) were worn for 2-3 minutes for EtCO2 and respiration assessments and physical fit assessment.
  Interventions: Device: Medline Pediatric Face Masks; Device: KC Childs Mask
- Children 10-12 yrs (Active Comparator): Medline Pediatric Face Mask KC Childs Face Mask
  Comparison of Medline Pediatric Face Masks and KC Childs Mask which are both single use disposable masks. Each mask (two in total) were worn for 2-3 minutes for EtCO2 and respiration assessments and physical fit assessment.
  Interventions: Device: Medline Pediatric Face Masks; Device: KC Childs Mask

INTERVENTIONS:
Device: Medline Pediatric Face Masks — Medline Face Masks, which are single use disposable masks were evaluated on children. The mask was worn for 2-3 minutes for EtCO2 and respiration assessments and physical fit assessment.
Device: KC Childs Mask — KC Childs Mask, which are single use disposable masks were evaluated on children. The mask was worn for 2-3 minutes for EtCO2 and respiration assessments and physical fit assessment.

SUMMARY:
Compare the fit of two pediatric face masks in children.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label comparative observational study to be conducted in up to two (2) facilities with the healthy and non-healthy Subjects (4-12 years of age). The usage of face masks is common practice within hospitals, and masks may be evaluated outside of clinical facilities as well.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 12 years of age
* conscious

Exclusion Criteria:

* able to wear a mask
* no previous allergic reactions to face masks

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Drower, MS, Principal Investigator — Medline Industries, Inc
Locations (1):
- Medline Industries, Inc, Mundelein, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Statistical analysis projected ninety-nine (99) Subjects were needed to assess mask equivalence, however only 96 subjects were enrolled at the facility.
Groups:
- Medline Face Mask First: Medline Face Mask first, then KC Childs Mask
- KC Childs Mask First: KC Childs Mask first, then Medline Face Mask
Period: Overall Study
Arm/Group | Medline Face Mask First | KC Childs Mask First
Started | 48 | 48
Completed | 48 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Partipants: All subjects were randomized to all interventions -- Medline Pediatric Face Mask and KC Childs
Arm/Group | All Study Partipants
Number analyzed (Participants) | 96
Age, Customized [Count of Participants; unit: Participants]
  4-5 years | 19
  6-9 years | 45
  10-12 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 96
EtCO2 [Mean (Standard Deviation); unit: mmHg]
  Medline Mask | 40.7 (4.4)
  KC Mask | 40.8 (4.3)
Respiration Rate [Mean (Standard Deviation); unit: breaths per minute]
  Medline Mask | 19.3 (3.4)
  KC Mask | 19.0 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Carbon Dioxide Levels
Description: ETCO2 will be assessed by a capnographer when wearing each pediatric face mask. Results are the difference between masks in change from baseline.
Time Frame: Baseline and 2 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Medline Pediatric Face Mask: All participants Medline Pediatric Face Mask
- KC Childs Mask: All subjects KC Childs Mask
Arm/Group | Medline Pediatric Face Mask | KC Childs Mask
Number analyzed (Participants) | 96 | 96
mmHg | -0.07 (3.56) | -0.79 (0.65)

2. Secondary Outcome: Physical Fit of Pediatric Face Masks.
Description: Physical fit will be determined by a reviewer after the mask is put on. The fit will be based on a several fit parameters to compare the difference in the score between the two masks.
  The total fit score was calculated by summing the nose to chine coverage score (0 = No, 1=Yes) and gap score (0=No apparent gap, flush to face on one or both sides, 1=Slight gap, not flush to face but can see cheeks only, 2=Moderate gap, can see mouth. , 3=Large gap, mask loose fitting all around face (chin, sides, nose, etc.) to arrive a total score with 0 indicating best fit and 4 indicating worst fit.
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Particpants: Medline Pediatric Face Mask KC Childs Face Mask
Arm/Group | All Particpants
Number analyzed (Participants) | 96
units on a scale
  Medline Mask | .80 (.79)
  KC Mask | .31 (.59)

3. Other Pre Specified Outcome: Change From Baseline in Respiration Rates
Description: Change from Baseline
Time Frame: Baseline and 2 minutes
Population: Respiration Rate
Measure: Mean (Standard Deviation); unit: Breaths per minute
Groups:
- All Participants: Medline Pediatric Face Mask KC Childs Face Mask
Arm/Group | All Participants
Number analyzed (Participants) | 96
Breaths per minute
  Medline Mask | -1.14 (.41)
  KC Mask | -1.0 (2.8)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Medline Pediatric Face Mask: Medline Face Mask
- KC Childs Face Mask: KC Face Mask
Arm/Group | Medline Pediatric Face Mask | KC Childs Face Mask
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/96
Other Adverse Events (participants affected / at risk) | 0/96 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No